CLINICAL TRIAL: NCT05705947
Title: Patient Reported Outcomes Following Low-dose Irradiation for Osteoarthritis (PRO-LO): A Single-arm Prospective Registry
Brief Title: PROs Following Low-dose Irradiation for Osteoarthritis
Acronym: PRO-LO
Status: Active, not recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 22-3256
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; radiation therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with osteoarthritis receiving radiation treatment: Patients with osteoarthritis receiving standard of care radiation treatment at UNC Radiation Oncology clinic. Radiation dose and fractionation prescription is at the physician's discretion.
  Typically, this prescription is delivered in 6 fractions, every other day, over 2 weeks.

SUMMARY:
The goal of this observational registry study is to collect data related to patient reported outcomes (pain, function, quality of life, toxicity) in osteoarthritis (OA) patients receiving standard of care radiation therapy (RT).

DETAILED DESCRIPTION:
This is a single-institution, single-arm, prospective, observational study of patients with osteoarthritis who are being treated with standard of care radiation therapy (RT). The purpose of this non-interventional study is to systematically collect data related to patient reported outcomes (pain, function, quality of life, toxicity) with the goal of optimizing approaches to management with radiation therapy and clinical care during follow up. The primary endpoint of this study is a change in visual analog pain scale (VAPS) at 3 months post radiation and a variety of secondary endpoints are aimed at assessing disease control, patient function, avoidance of invasive surgery, and toxicity. Participants will complete patient-reported outcome surveys for pain and joint-specific functional assessment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Established diagnosis of OA of at least 1 joint
* Inadequately controlled pain due to OA despite attempts with 2 or more other treatment modalities and Visual Analogue Pain Score of 4 or greater.
* Will undergo radiation as part of their standard of care for OA.
* At least 55 years old
* Ability to read and speak English.

Exclusion Criteria:

* Any woman who is pregnant or has reason to believe she is pregnant (the possibility of pregnancy has to be excluded by negative urine ß-HCG results, obtained within 2 weeks of CT simulation for radiation planning, or on the basis of patient history, e.g.: tubal ligation, hysterectomy or a minimum of 1 year without menses).
* Estimated life expectancy less than 6 months.
* Radiation treatment for shoulder OA
* Patient weight greater than 550lbs

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged 55 or above, who are receiving radiation treatment at UNC Radiation Oncology for Osteoarthritis are the intended study population.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Pain Scale (VAPS) Score from Baseline to M3 Post Radiation Treatment Completion | Baseline and 3 months post RT
  The investigators will use the visual analog 0-10 pain scale (VAPS) and compare the baseline pre-radiation measurement to that measured at 3 months post radiation.

SECONDARY OUTCOMES:
Change in Visual Analog Pain Scale (VAPS) Score Over Time | Baseline up to 5 years post RT
  The investigators will use the visual analog 0-10 pain scale (VAPS), where 0 is no pain and 10 is the worst physical pain imaginable, and compare the baseline pre-radiation measurement to that assessed at 6 weeks, 6 and 12 months, and yearly up to 5 years post radiation (RT). Higher scores indicate a worse outcome.
Change in Hip Joint-Specific Outcome Over Time | Baseline up to 5 years post RT
  Joint-specific outcomes measures scales will include the Hip Injury and Osteoarthritis Outcome Score (HOOS). With 1 being the most functional usage of the joint, and 5 being least functional usage of the joint. The higher the value, the less functional outcome of the joint. Investigators will compare the baseline pre-radiation measurement to that assessed at 6 weeks, 3, 6 and 12 months, and yearly up to 5 years post radiation.
Change in Knee Joint-Specific Outcome Over Time | Baseline up to 5 years post RT
  Joint-specific outcomes measures scales will include the Knee Injury and Osteoarthritis Outcome Score (KOOS). With 1 being the most functional usage of the joint, and 5 being least functional usage of the joint. The higher the value, the less functional outcome of the joint. It will compare the baseline pre-radiation measurement to that assessed at 6 weeks, 3, 6 and 12 months, and yearly up to 5 years post radiation.
Change in Arm, Shoulder and Hand Joint-Specific Outcome Over Time | Baseline up to 5 years post RT
  Joint-specific outcomes measures scales will include the Disability of Arm Shoulder and Hand (DASH). With 1 being the most functional usage of the joint, and 5 being least functional usage of the joint. The higher the value, the less functional outcome of the joint. It will compare the baseline pre-radiation measurement to that assessed at 6 weeks, 3, 6 and 12 months, and yearly up to 5 years post radiation.
Change in Foot Joint-Specific Outcome Over Time | Baseline up to 5 years post RT
  Joint-specific outcomes measures scales will include the Foot & Ankle Disability Index Score (FADI). With 1 being the most functional usage of the joint, and 5 being least functional usage of the joint. The higher the value, the less functional outcome of the joint. It will compare the baseline pre-radiation measurement to that assessed at 6 weeks, 3, 6 and 12 months, and yearly up to 5 years post radiation.
Change in NSAID Dosage | Baseline up to 5 years post RT
  The investigator will compare NSAID doses at baseline to that measured at 6 weeks, 3, 6, and 12 months, and yearly up to 5 years post-radiation.
Change in Opioid Dosage | Baseline up to 5 years post RT
  The investigator will compare opioid doses at baseline to that measured at 6 weeks, 3, 6, and 12 months, and yearly up to 5 years post-radiation.
Change in NSAID Frequency | Baseline up to 5 years post RT
  The investigator will compare NSAID frequencies at baseline to that measured at 6 weeks, 3, 6, and 12 months, and yearly up to 5 years post radiation.
Change in Opioid Frequency | Baseline up to 5 years post RT
  The investigator will compare opioid frequencies at baseline to that measured at 6 weeks, 3, 6, and 12 months, and yearly up to 5 years post radiation.
Invasive Procedures | Up to 5 years post RT
  The investigator will report invasive procedures to treat the radiated joint experienced by each subject for the treatment of OA.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Yanagihara, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No